CLINICAL TRIAL: NCT05508217
Title: Impact of Telomere Biology and Sperm DNA Fragmentation on Embryonic Development
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: IVI Madrid (Other)
Responsible Party: Sponsor
Other Study IDs: 2202-MAD-024-CB
Record Dates: First submitted 2022-08-16; First posted 2022-08-19 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2024-01

CONDITIONS: Sperm DNA Fragmentation; Male Fertility; Telomeres; Sperm
Keywords: Sperm DNA fragmentation; Telomeres; Sperm; Male fertility; Sperm telomeric length

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Semen samples will be obtained on the day of oocyte fertilization and the unused part of the sample is recovered for Sperm LT determination, ST accumulation, sperm DNA fragmentation and sperm maturation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The proposed project we intend to assess the implication of the telomeric pathway in male infertility. To get this, several analyzes will be carried out: 1. Determination of the TL by means of two methods: Q-FISH and PCR. 2. Determination of sperm DNA fragmentation by tunnel technique. 3. Assess sperm maturation.

Finally, the correlations between age, normality or not of the seminogram, LT, Short telomers (ST) accumulation, DNA fragmentation levels, sperm maturation and fertility, blastocyst development, and pregnancy rates will be established in search of cut-off points that can give a forecast of man´s fertility who consults on this subject.

DETAILED DESCRIPTION:
To carry out the project, men who come to the clinic in the context of a couple fertility study and who do not have a known cause that justifies their infertility will be recruited. A clinical history will be made, and an informed consent will be given to them for their participation in the project (Annex Consents). Semen samples will be obtained on the day of oocyte fertilization and the unused part of the sample is recovered for Sperm LT determination, ST accumulation, sperm DNA fragmentation and sperm maturation.

ELIGIBILITY:
Inclusion Criteria:

* Men of any age who come to IVI Madrid in the context of a couple's infertility study and who present normozoospermia or semenograms with sperm count >10mill/ml, >25% progressive motility and > 1% normal morphology.

Exclusion Criteria:

* Males who have suffered any acute illness in the three months prior to inclusion in the study.
* Males with any known chronic disease or genetic alteration.

Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Men of any age who come to IVI Madrid in the context of a couple's infertility study and who present normozoospermia or semenograms with sperm count >10mill/ml, >25% progressive motility and > 1% normal morphology.
Study Population: The target population is men with normozoospermia attending the IVI Madrid clinic. Men with oligoasthenozoospermic subfertility will also be taken in order to compare data with more extreme situations. However, the results of the study (a possible telomeric length and DNA fragmentation analysis kit) are intended to be applied to normozoospermic men whose infertility is classified as idiopathic, i.e. despite normal laboratory results, no cause for their reproductive problem can be found.
  Translated with www.DeepL.com/Translator (free version)
Sampling Method: Non-Probability Sample
Enrollment: 204 (Estimated)
Dates: Start 2022-08-22 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
To assess the correlation between the length of the telomeres of the spermatozoa used in ICSI treatments with donor oocytes and their rate of blastocyst development. | 6 months
  Characterisation of telomeric factors (telomere length, percentage of short telomeres, DNA damage) in men undergoing fertility treatments using donor oocytes, in order to find out whether telomeric parameters can be a predictive factor for fertility.

SECONDARY OUTCOMES:
Methods of telomere measurement PCR and Q-FISH will be evaluated in order to assess whether the results are superimposable and to determine their advantages and disadvantages. | 6 months
  With the proposed project we intend to assess the implication of the telomeric pathway in male infertility. To get this, several analyzes will be carried out:
  1. Determination of the TL by means of two methods: Q-FISH and PCR.
Methods of telomere measurement PCR and Q-FISH will be evaluated in order to assess whether the results are superimposable and to determine their advantages and disadvantages. | 6 months
  With the proposed project we intend to assess the implication of the telomeric pathway in male infertility. To get this, several analyzes will be carried out:
  2. Determination of sperm DNA fragmentation by tunnel technique.
Methods of telomere measurement PCR and Q-FISH will be evaluated in order to assess whether the results are superimposable and to determine their advantages and disadvantages. | 6 months
  With the proposed project we intend to assess the implication of the telomeric pathway in male infertility. To get this, several analyzes will be carried out:
  3. Assess sperm maturation.
Percentage of short telomeres in samples analysed by FISH will be establish. | 6 months
  To establish the percentage de short telomeres in the samples to know a new biomark.
To determine the sperm DNA fragmentation measured by Tunel assay and its correlation with the rate of blastocyst development. | 6 months
  To establish the relationship of DNA fragmentation and the blastocyst development
Correlation of telomere length data with sperm DNA fragmentation levels, as well as fertilization, implantation, blastocyst development and pregnancy rate and live-birth. | 6 months
  To know the important of telomere length and DNA fragmentation levels for sucessful treatment
To assess if there is a correlation between embryo morphokinetic parameters and telomere length, levels of sperm DNA fragmentation, BMI and paternal age. | 6 months
  To know the male characteristics that influence the treatment
Establish an algorithm on the degree of male fertility based on different combinations with the previously collected data: telomere length, sperm DNA fragmentation, fertilization rates, blastocyst formation rate, pregnancy and live newborn. | 6 months
  To know the male characteristics that influence the treatment

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Balmori Boticario, PhD, Principal Investigator — IVI Madrid
Locations (1):
- Ivirma Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No